CLINICAL TRIAL: NCT05856994
Title: Clinical Assessment of Protopic® Ointment in Deep Partial-Thickness Burns
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wesley Thayer, Clinical Professor of Plastic Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 222242
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Burn Injury
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tacrolimus Ointment 0.03% with hydrocolloid dressing (Experimental): Standard out-patient wound cleaning followed by application of tacrolimus ointment over the burn and hydrocolloid dressing on the treated area.
  Interventions: Drug: Tacrolimus ointment
- Bacitracin ointment (No Intervention): Standard out-patient wound cleaning followed by application of bacitracin ointment over the burn and hydrocolloid dressing on the treated area.
- Hydrocolloid dressing (No Intervention): Standard out-patient wound cleaning followed by application of hydrocolloid dressing on the burned area.

INTERVENTIONS:
Drug: Tacrolimus ointment — For the active comparator group, the wound(s) will be cleaned and bacitracin ointment will be applied to the wound. External dressings on all treated wounds will be placed based on the current standard of care. For the control group, the wound(s) will be cleaned and a hydrocolloid Dressing will be affixed to the burn and treated area. For the treatment group, the wound(s) will be cleaned and tacrolimus (0.03%) ointment will be applied over the burn. Hydrocolloid Dressing will be affixed to the burn and treated area. External dressings on all treated wounds will be placed based on the current standard of care.
  Other Names: Protopic® ointment
  Arms: Tacrolimus Ointment 0.03% with hydrocolloid dressing

SUMMARY:
There is currently no standard treatment to prevent burn depth conversion in partial-thickness burns. Conversion into deeper wounds is associated with higher complications and morbidity. The most common theory attributes this depth conversion to the prolonged inflammatory response that occurs after burn injury. Therefore, the investigators propose testing the safety and efficacy of tacrolimus ointment (an immunosuppressive agent) in patients with deep partial-thickness burns.

DETAILED DESCRIPTION:
Patients who sustain burn injuries are some of the most complex patients to care for, often requiring a multidisciplinary team of providers specialized in burn pathophysiology. While many facets of burn care must be accounted for including fluid management, nutrition, respiratory status, immunologic and cardiovascular function, innovation in the treatment for deep partial thickness burns is of paramount importance.

Burn depth conversion is a phenomenon where superficial partial-thickness burns spontaneously convert into deep partial-thickness or full-thickness burns, which are associated with higher complications and morbidity. The most common theory attributes this depth conversion to the prolonged inflammatory response that occurs after burn injury. Excess inflammation worsens the injury through various mechanisms, including cytokine production, delayed inflammatory cell apoptosis, and reactive oxidative species production.

Protopic® (tacrolimus) Ointment is a macrolide immunosuppressant and a calcineurin inhibitor. Tacrolimus inhibits T-lymphocyte activation, a key cell in the body's immune response. A prolonged inflammatory response is theorized to contribute to a worse recovery outcome in partial- to full-thickness burns. Therefore, tacrolimus possesses properties that could slow the acute inflammatory response and potentially improve clinical outcomes in deep partial-thickness burns. There has yet to be a clinical study to investigate the use of tacrolimus in burn treatment. However, our group recently published an animal study that found a significant reduction in burn depth using tacrolimus topically (White-Dzuro et al. Burns 2022). This study is a randomized clinical trial of the usage of tacrolimus ointment for the treatment of deep partial-thickness burns with comprehensive assessments of healing and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form by the subject or Legally Authorized Representative.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female aged 50 to 75 at time of screening visit.
* For females of reproductive potential, confirmed negative urine pregnancy test at enrollment.
* Presence of deep partial-thickness burns to one or both dorsal hands (burns may be present on other areas of the body, so long as all regions combined are ≤ 5% Total Body Surface Area [TBSA], using the Browder and Lund Chart).
* Thermal burn (caused by fire, hot objects, steam or hot liquids [scalding]) etiology, located on one or both dorsal hands.
* Ability to implement treatment within 24-48 hours days of the initial burn.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study, if applicable.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Allergy or hypersensitivity to tacrolimus or other components of the ointment (per subject report) or personal preference.
* Allergy or hypersensitivity to bacitracin and/or any of its drug formulation components. Patients with known hypersensitivity to neomycin may also be sensitive to bacitracin.
* Subject is incarcerated.
* Friction, chemical or electric burn etiology.
* Immunosuppression, as determined by the Principal Investigator.
* Presence of a local and/or systemic infection that, in the Investigator's opinion, requires aggressive treatment which would warrant exclusion from participating in this study.
* Subject is unwilling or unable to follow study related procedures and/or follow-up visits.
* Prior treatment to the burn wound(s) on the hand(s) considered for this trial with another product (treatment failure).
* Subject report of previous participation in another interventional burn wound study within 60 days prior to the Screening Visit.
* Subject report of concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
* The subject has any physical or psychiatric condition that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete wound healing | 21 days
  Clinical burn wound assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Thayer, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No